CLINICAL TRIAL: NCT00256295
Title: A Phase II Study of Weekly Oxaliplatin and Gemcitabine Combination Chemotherapy for Recurrent or Metastatic Head and Neck Cancer
Brief Title: Weekly Oxaliplatin and Gemcitabine for Recurrent or Metastatic Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sai-Hong Ignatius Ou (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Sai-Hong Ignatius Ou, Dr. Sai-Hong Ignatius Ou, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 04-08; 2004-3776 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Cancer of the Head and Neck
Keywords: Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine plus Oxaliplatin (Experimental): Gemcitabine given 1000 mg/m2 IV over 100 minutes Every 21 days. Oxaliplatin given 65 mg/m2 IV over 120 minutes immediately following gemcitabine Every 21 days.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 IV over 100 minutes Every 21 days
  Other Names: Gemzar; NSC-613327
Drug: Oxaliplatin — 65 mg/m2 IV over 120 minutes immediately following gemcitabine Every 21 days
  Other Names: NSC-266046

SUMMARY:
The combination of oxaliplatin and gemcitabine is highly active in a wide variety of tumors including pancreatic, germ cell, breast, biliary, mesothelioma (Mitchell et al, 2002), and lung. In the last study which utilized days 1 and 8 gemcitabine 1000 mg/m2 and days 1 and 8 oxaliplatin 65 mg/m2 in poor prognosis lung cancer patients (PS 1-3) the response rate was 16% with no incidence of febrile neutropenia.

Toxicity is a crucial consideration when designing regimens intended for palliation. Toxicities associated with cisplatin can make it difficult to use in patients with Head and Neck Cancer (HNC), many of whom are elderly and have comorbidities. In addition, many patients with metastatic HNC have previously received cisplatin during neoadjuvant/adjuvant therapy, or as part of their primary chemoradiation treatment. When these patients recur, it is possible their tumors have innate or acquired cisplatin resistance. Oxaliplatin is likely to be better tolerated than cisplatin containing regimens, especially with regards to neurotoxicity. Gemcitabine has shown promising activity as a single agent and in combination chemotherapy in the first line treatment of patients with HNC. A combination chemotherapy regimen using oxaliplatin and gemcitabine administered once every week is logical and worth exploring in patients with metastatic and recurrent head and neck cancer to improve the toxicity profile and patient monitoring while maintaining efficacy of the chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck region. Primary tumor sites include: lip, oral cavity, pharynx (oropharynx, hypopharynx), or larynx (supraglottis, glottis, subglottis). For nasopharynx primary, all squamous histologic subtypes are allowed (WHO type-I keratinizing, WHO type-II non-keratinizing, WHO type-III undifferentiated).
* Patients must have metastatic or locally recurrent carcinoma of the head and neck. Patients with locoregional disease must be considered incurable by means of locoregional therapy.
* All sites of disease must be assessed and designated as measurable or non-measurable disease as documented by CT, MRI, X-ray physical exam or nuclear exam. All measurable disease must be assessed within 28 days prior to registration. All non-measurable disease must be assessed within 42 days prior to registration.
* Patients may have received prior radiotherapy if there has been complete recovery from all radiation-induced toxicities. At least 4 weeks must have been elapsed from the completion of radiation therapy to the time of registration. If lesions within the radiation port are to be used to assess response to therapy, those lesions must have demonstrated clear progression following completion of radiation therapy.
* Patients must have adequate bone marrow reserve as documented by absolute neutrophil count (ANC) > 1,500 microliters and platelets > 100,000/microliter obtained within 14 days prior to registration.
* Patients must have adequate hepatic as documented by serum bilirubin < 1.5 x the institutional upper limit of normal. Serum transaminase (SGOT or SGPT) must be < 1.5 x the institutional upper limit of normal serum unless the liver is involved with tumor, in which case serum transaminase (SGOT or SGPT) must be < 5 x the institutional limit of normal. These tests must be obtained within 14 days prior to registration.
* Patients must have a creatinine < 1.5 x the institutional upper limit of normal or a creatinine clearance of > 30 cc/min calculated using the following formula obtained within 28 days prior to registration.

Calculated Creatinine Clearance = (140-age) X wt (kg) X (0.85 if female) 72 X creatinine (mg/dl)

These tests must have been performed within 28 days prior to registration.

* All patients must be 18 years of age or older
* Patients must have a Zubrod performance of 0-2

Exclusion Criteria:

* Patients must not have more than one prior chemotherapy regimen for recurrent/metastatic disease. Patients with initial locally advanced but non-metastatic disease are allowed to have one prior chemotherapy regimen as part of the primary curative therapy. All chemotherapy must be completed 4 weeks prior to registration. Any number of prior biologic therapies (e.g. chimeric antibodies or kinase inhibitors) is permitted as part of the chemotherapy regimen.
* Patients must not have a surgical treatment procedure for head and neck cancer within 4 weeks prior to registration. Surgical procedure for biopsy purpose alone is allowed within 28 days prior to registration. Patients must have completely recovered from all surgery prior to registration.
* Patients must not have prior therapy with oxaliplatin or gemcitabine
* Patients with any evidence of active or uncontrolled infection, recent myocardial infection, unstable angina, or life threatening arrhythmia are not eligible.
* Patients with severe psychiatric disorder are not eligible.
* Patients with known brain metastasis are not eligible. However, brain-imaging studies are not required for eligibility if the patient has no neurological signs or symptoms. If brain-imaging studies are performed, they must be negative for disease.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell carcinoma, in situ cervical cancer, or adequately treated Stage I and II cancer from which the patient is in complete remission, or any other malignancy from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-04; Primary Completion 2008-02 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignatius Ou, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: April 2005 Primary completion date: February 2008 Study completion date: October 2011
Groups:
- Gemcitabine Plus Oxaliplatin: Gemcitabine given 1000 mg/m2 IV over 100 minutes Every 21 days. Oxaliplatin given 65 mg/m2 IV over 120 minutes immediately following gemcitabine Every 21 days.
  Gemcitabine : 1000 mg/m2 IV over 100 minutes Every 21 days
  Oxaliplatin : 65 mg/m2 IV over 120 minutes immediately following gemcitabine Every 21 days
Period: Overall Study
Arm/Group | Gemcitabine Plus Oxaliplatin
Started | 7 (Of the 8 subjects consented, 1 withdrew prior to treatment.)
Completed | 3
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine Plus Oxaliplatin
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Response)
Description: Complete Response (CR): Complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. Normalization of markers and other abnormal lab values. All disease must be assessed using the same techniques as baseline.
  Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: 5 years
Population: No subject data were analyzed; therefore, data cannot be summarized for inclusion in these data tables.
Arm/Group | Gemcitabine Plus Oxaliplatin
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency and Severity of Toxicities
Time Frame: 5 years
Population: No subject data were analyzed; therefore, data cannot be summarized for inclusion in these data tables.
Arm/Group | Gemcitabine Plus Oxaliplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival and Time to Treatment Failure
Time Frame: 5 years
Population: No subject data were analyzed; therefore, data cannot be summarized for inclusion in these data tables.
Arm/Group | Gemcitabine Plus Oxaliplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Gemcitabine Plus Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Plus Oxaliplatin (N=7)
Death due to disease progression (General disorders) | 4 (4) — These events were not study related.
Dehydration due to disease progression (Metabolism and nutrition disorders) | 1 (1) — This event was not study related.
Pneumonia due to disease progression (Infections and infestations) | 1 (1) — This event was not study related.
Carotid artery rupture due to disease progression (Vascular disorders) | 1 (1) — This event was not study related.
Grade II Hepatic toxicity (Hepatobiliary disorders) | 1 (1) — This event was not study related.
Broken leg due to fall (General disorders) | 1 (1) — This event required hospitalization and was not study related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine Plus Oxaliplatin (N=7)
Grade 3 Sinus Tachycardia (Cardiac disorders) | 1 (1) — This event was not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes